CLINICAL TRIAL: NCT05155852
Title: NIRS-Based Bedside Monitoring to Identify Impaired Cerebral Autoregulation in Women with Postpartum Hypertension
Brief Title: Bedside Monitoring to Identify Impaired Cerebral Autoregulation in Women with Postpartum Hypertension
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Eliza Miller MD MS, Assistant Professor of Neurology in the Division of Stroke and Cerebrovascular Disease, Columbia University
Other Study IDs: AAAT1562; 3K23NS107645-02S1 (NIH)
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Preeclampsia; Hypertension in Pregnancy
Keywords: Near-infrared spectroscopy (NIRS); Preeclampsia; Pregnancy
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Post-delivery preeclampsia patients: Women admitted to the high-risk unit(s) with elevated blood pressure and neurological symptoms, such as headache, after delivery.

SUMMARY:
The purpose of this research study is to develop a protocol for NIRS-based bedside monitoring to identify impaired cerebral autoregulation in women admitted to the high-risk obstetrics unit with postpartum hypertension. The investigators will then pilot this protocol in 10 patients with high-risk neurological features, such as headache.

DETAILED DESCRIPTION:
Maternal neurological complications are a leading cause of postpartum severe maternal morbidity and maternal mortality (SMM/MM). The lack of biomarkers to identify women at highest risk of these rare, but devastating postpartum complications, including stroke, seizures, and posterior reversible encephalopathy syndrome, has impeded efforts to prevent neurological SMM/MM.

Impaired cerebral autoregulation may be such a biomarker. Preliminary results using transcranial Doppler (TCD) based techniques to quantify cerebral autoregulation have demonstrated severely impaired cerebral autoregulation in the postpartum period in some women. However, TCD is operator dependent, and cannot be used for extended monitoring due to discomfort. In contrast, near-infrared spectroscopy (NIRS) is fully automated and can be continued for hours at the bedside. Identifying personalized blood pressure (BP) targets using NIRS has been shown to improve outcomes in acute stroke patients, another population with impaired cerebral autoregulation. However, this method has not been applied in postpartum women.

This is a single center feasibility study that will include up to 10 women. Postpartum women admitted to the obstetrics high-risk stepdown unit for management of postpartum hypertension will be eligible for this study. Informed consent will be obtained from participants prior to enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* Women who have given birth within the previous 12 weeks
* Admitted to the high-risk inpatient obstetrics unit for management of hypertension
* With headache or other neurological symptoms such as vision changes

Exclusion Criteria:

* Acute ischemic stroke
* Intracerebral or subarachnoid hemorrhage
* Eclamptic seizures
* Any other neurological complication requiring transfer to the neurological intensive care unit or stroke stepdown unit
* History of Reynaud's syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from the high-risk inpatient obstetrics unit at NewYork-Presbyterian Hospital/Columbia University Irving Medical Center. Women who have given birth within the previous 12 weeks and are admitted to the high-risk inpatient obstetrics unit for management of hypertension will be screened.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Oxygenated hemoglobin concentration | Continuously collected for up to 24 hours
  The Edwards HemoSphere system with ForeSight Elite NIRS component (Edwards LifeSciences) will be used to monitor oxygenated and deoxygenated hemoglobin concentrations. Two adhesive NIRS probes will be placed on the frontotemporal scalp covering the cortex, usually supplied by the middle cerebral artery.
  [Describe how the concentration will be obtained, the range of anticipated concentrations, and how to interpret the concentrations - eg, higher concentrations indicate ...]
Deoxygenated hemoglobin concentration | Continuously collected for up to 24 hours
  The Edwards HemoSphere system with ForeSight Elite NIRS component (Edwards LifeSciences) will be used to monitor oxygenated and deoxygenated hemoglobin concentrations. Two adhesive NIRS probes will be placed on the frontotemporal scalp covering the cortex, usually supplied by the middle cerebral artery.
Blood pressure (BP) | Continuously collected for up to 24 hours
  Continuous non-invasive BP monitoring will be utilized (ClearSight finger cuff system, Edwards LifeSciences).

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Miller, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital (NYP), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersen NH, Silverman A, Strander SM, Kodali S, Wang A, Sansing LH, Schindler JL, Falcone GJ, Gilmore EJ, Jasne AS, Cord B, Hebert RM, Johnson M, Matouk CC, Sheth KN. Fixed Compared With Autoregulation-Oriented Blood Pressure Thresholds After Mechanical Thrombectomy for Ischemic Stroke. Stroke. 2020 Mar;51(3):914-921. doi: 10.1161/STROKEAHA.119.026596. Epub 2020 Feb 12. PMID 32078493